CLINICAL TRIAL: NCT05419388
Title: A Randomized, Open-Label, Multicenter, Phase II Study of Multiple Doses of RO7247669 in Participants With Previously Untreated Unresectable or Metastatic Melanoma
Brief Title: A Study of Multiple Doses of RO7247669 in Participants With Previously Untreated Unresectable or Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP43963; 2023-505672-30-00 (EU CTIS Number)
Record Dates: First submitted 2022-06-13; First posted 2022-06-15 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low dose every three weeks (Q3W) (Experimental): Participants will receive RO7247669 Q3W until loss of clinical benefit, unacceptable toxicity, or a maximum of 24 months.
  Interventions: Drug: RO7247669
- High dose Q3W (Experimental): Participants will receive RO7247669 Q3W until loss of clinical benefit, unacceptable toxicity, or a maximum of 24 months.
  Interventions: Drug: RO7247669

INTERVENTIONS:
Drug: RO7247669 — Participants will receive intravenous (IV) RO7247669 Q3W

SUMMARY:
The purpose of this study is to assess the efficacy, safety, pharmacokinetics (PK), and pharmacodynamics of two dose levels of RO7247669 in participants with unresectable or metastatic melanoma to select the recommended dose for further development.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable or metastatic melanoma, per the American Joint Committee on Cancer (AJCC) staging system (unresectable Stage III or Stage IV)
* Radiologically measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Known v-Raf murine sarcoma viral oncogene homolog B1 (BRAF) V600 mutation status
* Adequate cardiovascular, hematological, hepatic and renal function
* Willingness to abide by contraceptive measures for the duration of the study
* Participants must have known PD-L1 status

Exclusion Criteria:

* Pregnancy, lactation, or breastfeeding
* Known hypersensitivity to any of the components of RO7247669
* Participants must not have ocular melanoma
* Symptomatic central nervous system (CNS) metastases
* Significant cardiovascular/cerebrovascular disease within 6 months prior to randomization
* Known active or uncontrolled bacterial, viral, fungal, mycobacterial, parasitic, or other infection or any major episode of infection requiring treatment with intravenous (IV) antibiotics or hospitalization within 28 days prior to randomization
* Major surgical procedure or significant traumatic injury (excluding biopsies) within 28 days prior to randomization, or anticipation of the need for major surgery during the course of the study
* Active or history of autoimmune disease or immune deficiency with some exceptions
* Prior systemic anticancer therapy for unresectable or metastatic melanoma
* Prior anticancer therapy with any-immunomodulatory agents including CPIs (such as anti-programmed death-ligand 1[PD-L1]/PD-1 and anti-cytotoxic T lymphocyte-associated antigen [CTLA-4]) with some exceptions if used as prior adjuvant or neoadjuvant melanoma therapies
* Prior treatment with anti-LAG3 therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-11-27 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From randomization to the first occurrence of progression or death during the treatment period or within 60 days of the last tumor assessment after treatment discontinuation from any cause, whichever occurs first (up to 25 months)

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events | Up to 25 months
Objective response rate (ORR) | Up to 25 months
Disease control rate (DCR) | Up to 25 months
Duration of response (DOR) | From the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to 25 months)
Serum concentration of RO7247669 | Up to 25 months
Percentage of participants with anti-drug antibodies (ADAs) | Baseline up to 25 months
Change from baseline in the number and activation status of peripheral blood immune cells | Baseline up to 25 months
Change from baseline in the number and activation of immune cells in the tumor microenvironment | Baseline to Cycle 2 Day 9 (cycle = 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- Australia (4):
  - Coffs Harbour Health Campus, Coffs Harbour, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - One Clinical Research, Nedlands, Western Australia
- Brazil (4):
  - Hospital de Clínicas de Porto Alegre X, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- Všeobecná fakultní nemocnice v Praze, Prague, Czechia
- District General Hospital of Athens Laiko, Athens, Greece
- New Zealand (2):
  - Auckland City Hospital, Cancer and Blood Research, Auckland
  - Wellington Hospital, Wellington
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Narodowy Instytut Onkologii im. M.Sklodowskiej-Curie, Warsaw
- Slovakia (2):
  - Narodny Onkologicky Ustav, Bratislava
  - POKO Poprad, Poprad
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial, Barcelona
- Turkey (Türkiye) (3):
  - Adana Baskent University Hospital, Adana
  - Memorial Ankara Hastanesi, Ankara
  - Medipol Mega Üniversite Hastanesi Göztepe, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing